CLINICAL TRIAL: NCT04745832
Title: A Phase 3, Randomized, Open-Label, Controlled, Multicenter Study of Zandelisib (ME- 401) in Combination With Rituximab Versus Standard Immunochemotherapy in Patients With Relapsed Indolent Non Hodgkin's Lymphoma (iNHL) - The COASTAL Study
Brief Title: Phase 3 Study of Zandelisib (ME-401) in Combination With Rituximab in Patients With iNHL - (COASTAL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinuation of zandelisib program
Sponsor: MEI Pharma, Inc. (Industry)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME-401-004; 2020-004199-16 (EudraCT Number)
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2022-12

CONDITIONS: Follicular Lymphoma (FL); Non Hodgkin Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone | interventions — ME-401; Rituximab; Bendamustine Hydrochloride; Cyclophosphamide; Prednisone

STUDY DESIGN:
Intervention Model Description: Arm 1: Rituximab plus Zandelisib
  Arm 2: Rituximab plus chemotherapy (CHOP or Bendamustine)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rituximab plus Zandelisib (Experimental): Rituximab plus Zandelisib for 6 cycles followed by Zandelisib for 20 cycles
  Interventions: Drug: Zandelisib; Drug: Rituximab
- Rituximab plus chemotherapy (Experimental): Rituximab and Bendamustine or Rituximab with (CHOP) for 6 cycles
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: CHOP

INTERVENTIONS:
Drug: Zandelisib — Zandelisib 60 mg capsules taken daily for two cycles followed by intermittent schedule starting at Cycle 3
  Other Names: ME-401
  Arms: Rituximab plus Zandelisib
Drug: Rituximab — Rituximab IV 375 mg/m2 for 6 cycles
  Other Names: Rituxan; MabThera
Drug: Bendamustine — Bendamustine IV 90 mg/m2 on Days 1 and 2 for 6 cycles
  Other Names: Bendeka, Treanda, Belrapzo
  Arms: Rituximab plus chemotherapy
Drug: CHOP — Cyclophosphamide, Vindcristine IV, and Prednisone daily orally
  Other Names: cyclophosphamide 750 mg/m2, hydroxydoxorubicin IV 50 mg/m2, vincristine IV 1.4 mg/m2 and prednisone 100 mg daily
  Arms: Rituximab plus chemotherapy

SUMMARY:
This is a Phase 3 study of the PI3Kδ inhibitor Zandelisib (ME-401) in combination with rituximab, in comparison to standard immunochemotherapy (Rituximab-Bendamustine or Rituximab-CHOP) in subjects with relapsed or refractory FL and MZL.

DETAILED DESCRIPTION:
This is an open label, randomized, two-arm Phase 3 study in subjects with relapsed or refractory FL and MZL to evaluate efficacy and safety of zandelisib in combination with rituximab in comparison to standard immunochemotherapy (Rituximab-Bendamustine or Rituximab-CHOP).

Subjects must have relapsed after at least one previous line of systemic immunochemotherapy. Previous treatments must have included an anti-CD20 monoclonal antibody (mAb) with chemotherapy such as Bendamustine (B), CHOP, CVP, FND, or similar regimens, or an anti-CD20 mAb with Lenalidomide (L).

Approximately 534 randomized subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years of age, ≥19 years in Korea, or ≥20 years for subjects in Japan and Taiwan
* Histologically confirmed diagnosis of CD20 positive iNHL with histological subtype limited to:

  1. FL Gr 1, Gr 2, or Gr 3a
  2. MZL (splenic, nodal, or extra-nodal)
* Subjects with relapsed or refractory disease who received ≥1 prior lines of therapy
* Subjects must have at least one bi-dimensionally measurable lesion >1.5 cm
* Adequate hematologic parameters at screening unless abnormal values are due to disease
* Adequate renal and hepatic function
* Adequate cardiac function based on ECG and LVEF assessments

Exclusion Criteria:

* Histologically confirmed diagnosis of FL Gr 3b or transformed disease
* Prior therapy with PI3K inhibitors
* Ongoing or history of drug-induced pneumonitis
* Known lymphomatous involvement of the central nervous system
* Tested positive for or active viral infection with hepatitis B or C virus
* Tested positive or active infection with human immunodeficiency virus
* Tested positive, or active infection with human T-cell leukemia virus type 1
* Any uncontrolled clinically significant illness
* History of clinically significant cardiovascular abnormalities such as congestive heart failure
* History of clinically significant gastrointestinal (GI) conditions
* Females who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (141):
- United States (14):
  - The Oncology Institute of Hope and Innovation, Tucson, Arizona
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - The Oncology Institute of Hope and Innovation, Riverside, California
  - BRCR Medical Center Inc, Hollywood, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Revive Research Institute, Farmington Hills, Michigan
  - Revive Research Institute, Sterling Heights, Michigan
  - Mercy Clinic Cancer & Hematology - Chub O'Reilly Cancer Center, Springfield, Missouri
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - MetroHealth Medical Center, Cleveland, Ohio
  - Alpha Research Institute, LLC, Baytown, Texas
  - Valley Cancer Associates, Harlingen, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
- Australia (3):
  - Canberra Hospital, Garran
  - The Perth Blood Institute (PBI), West Perth
  - Westmead Hospital, Westmead
- Belgium (5):
  - AZ Sint-Jan Burgge-Oostende AV, Bruges
  - UZ Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Center Hospitalier de Jolimont, Haine-Saint-Paul
  - UZ Leuven Campus Gasthuisberg, Leuven
- Canada (3):
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie, Sherbrooke, Quebec
  - McGill University Health Centre, Québec
- France (9):
  - CHU Estaing. Service d'hématologie clinique et de thérapie cellulaire adulte,, Clermont-Ferrand
  - Centre Hospitalier De Dunkerque - Service d'hématologie, Le Mans
  - Centre Hospitalier du Mans, Le Mans
  - Centre Leon Berard, Lyon
  - Hôpital Saint-Louis, Paris
  - CHU de Bordeaux - Maladies Du Sang, Centre François Magendie, Pessac
  - Centre Henri Becquerel, Service d'Hematologie, Rouen
  - CHU de Tours, Hôpital Bretonneau Centre, Tours
  - Institut De Cancerologie Gustave Roussy, Villejuif
- Georgia (4):
  - LTD Israeli-Georgian Medical Research Clinic "Helsicore", Tbilisi
  - M. Zodelava Hematology Center, Tbilisi
  - J.S.C. K. Eristavi National Center of Experimental and Clinic, Tbilisi
  - LTD "Medinvest" Institute of Hematology and Transfusiology, Tbilisi
- Greece (4):
  - General Hospital of Athens "Laiko", Department of Haematology and Bone Marrow Transplantation, Athens
  - University General Hospital of Ioannina, Department of Haematology, Ioannina
  - University General Hospital of Patras "Panagia H. Voitheia", Pátrai
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Hungary (3):
  - Országos Onkológiai Intézet Gyógyszerterápiás Központ Hematológia és Lymphoma Osztály, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Belgyogyaszati Klinika, Debrecen
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz,, Nyíregyháza
- Italy (16):
  - SOC Oncologia Medica e dei Tumori Immunocorrelati, Aviano
  - UO di Ematologia "L.e A.Seragnoli" Policlinico Sant'Orsola Malpighi, Bologna
  - U.O. Ematologia, Azienda Ospedaliera S. Croce e Carle, Cuneo
  - U.O. Ematologia - Azienda Ospedaliero-Universitaria Careggi, Florence
  - U.O. Clinica Ematologica, Genova
  - SC Oncologia Medica, Meldola
  - UOC Ematologia, Presidio Ospedaliero Papardo, Messina
  - UO Ematologia 1 Azienda ULSS 3 Serenissima, Distertto del veneziano - Ospedale dell'Angelo di Mestre, Mestre
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Dipartimento di Oncoematologia, Unità Linfomi, Ospedale, Milan
  - Divisione Oncoematologia, Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Ospedali Riuniti Via Sofia, Palermo
  - UO Ematologia, Ospedale Civile S.Maria delle Croci, Ravenna
  - UO Ematologia, Ospedale Infermi di Rimini AUSL Romagna, Rimini
  - Istituti Fisioterapici Ospitalieri, Roma
  - S.C. Oncoematologia Azienda Ospedaliera Santa Maria, Terni
- Japan (25):
  - National Hospital Organization Nagoya Medical Center, Naka-ku, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Minami, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kagoshima University Hospital, Sakuragaoka, Kagoshima-Shi, Kagoshima
  - University Hospital Kyoto Prefectural University of Medicine, Kamigyō-ku, Kyoto
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Anjo Kosei Hospital, Aichi
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Aichi
  - Aomori Prefectural Central Hospital, Aomori
  - Chiba Cancer Center, Chiba
  - Kyushu University Hospital, Fukuoka
  - Chugoku Central Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Kyoto University Hospital, Kyoto
  - National University Corporation Tohoku University Hospital, Miyagi
  - Aichi Cancer Center Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Osaka University Hospital, Osaka
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Tokyo
  - Keio University Hospital, Tokyo
- Netherlands (2):
  - Albert Schweizer Ziekenhuis, Hematology Department, Dordrecht
  - Spaarne Gasthuis, Oncology Department, Hoofddorp
- New Zealand (2):
  - Canterbury District Health Board, Haematology Department, Christchurch
  - Dunedin Hospital, Southern Blood and Cancer Service, Dunedin
- Poland (4):
  - Klinika Hematologii, Szpital Uniwersytecki, Bydgoszcz
  - Pratia MCM Krakow, Krakow
  - ARS Medical - Szpital, Oddzial hematologiczny, Piła
  - Centrum Medyczne Pratia Poznan, Skorzewo
- Serbia (6):
  - University Clinical Center of Serbia, Clinic for Hematology, Belgrade
  - Zvezdara University Medical Center, Clinical department for Hematology and Oncology, Belgrade
  - Clinical Hospital Center "Zemun", Clinic for Internal Medicine, Department for Hematology, Belgrade
  - Oncology Institute of Vojvodina, Clinic for Internal Oncology, Kamenica
  - University Clinical Center Kragujevac, Clinic for Hematology, Kragujevac
  - Clinical Center of Vojvodina, Clinic for Hematology, Novi Sad
- South Korea (13):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A university Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Jeollyang
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul
  - Ewka Womans University Mokdong Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (9):
  - Hospital Universitario Quironsalud, Alcorcón, Madrid
  - Hospital Universitari Vall d'Hebron, Vall d'Hebron Institute of Oncology, Barcelona
  - Hospital Universitario Mútua Terrassa, Barcelona
  - Institut Catalá d'Oncologia, Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Hospitalario de Navarra, Navarro
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Tainan
- Turkey (Türkiye) (6):
  - Gazi University Health Research and Application Hospital, Hematology Department, Ankara
  - Istanbul University Istanbul Medical Faculty, Hematology Department, Istanbul
  - Erciyes University Medical Faculty, Department of Hematology, Kayseri
  - Ondokuz Mayis University Medical Faculty, Hematology Department, Samsun
  - Namik Kemal University Hospital, Tekirdağ
  - Karadeniz Technical University Medical Faculty Department of Hematology, Trabzon
- United Kingdom (9):
  - North Wales Cancer Treatment Centre, Bodelwyddan, Denbighshire
  - Royal Cornwall Hospital, Cornwell
  - Department of Haematology St. George's University of London, London
  - The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital, London
  - Imperial College Healthcare NHS Trust Hammersmith Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Genesis Care Oxford, Oxford
  - University Hospitals Plymouth NHS Trust, Derriford Hopital, Plymouth
  - The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital, Surrey Quays

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open from August 2021 through March 2023 at 144 investigational sites in the US, Argentina, Australia, Belgium, Canada, Czech Republic France Georgia, Germany, Greece, Hungary, Ireland, Italy, Japan, Korea, Netherlands, Poland, Serbia, Spain, Taiwan, Turkey, and UK
  Originally, it was anticipated that approximately 534 subjects would be randomized into the study however the study was terminated for business reasons with 82 subjects enrolled and dosed.
Groups:
- Rituximab Plus Zandelisib: Rituximab plus Zandelisib for 6 cycles followed by Zandelisib for 20 cycles Zandelisib: Zandelisib 60 mg capsules taken daily for two cycles followed by intermittent schedule starting at Cycle 3 Rituximab: Rituximab IV 375 mg/m2 for 6 cycles
  In the Rituximab plus Zandelisib arm, 41 subjects enrolled
- Rituximab Plus Chemotherapy: Rituximab and Bendamustine or Rituximab with (CHOP) for 6 cycles Rituximab: Rituximab IV 375 mg/m2 for 6 cycles Bendamustine: Bendamustine IV 90 mg/m2 on Days 1 and 2 for 6 cycles CHOP: Cyclophosphamide, Vindcristine IV, and Prednisone daily orally
  In the R-chemo arm 31 subjects were enrolled to R-B and 10 to R=CHOP
Period: Overall Study
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 21 | 21 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 18 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 0 | 1
  United States | 0 | 1 | 1
  Japan | 10 | 7 | 17
  United Kingdom | 4 | 2 | 6
  Spain | 0 | 1 | 1
  New Zealand | 0 | 1 | 1
  Netherlands | 1 | 0 | 1
  South Korea | 5 | 10 | 15
  Turkey | 1 | 3 | 4
  Belgium | 3 | 1 | 4
  Taiwan | 1 | 1 | 2
  Poland | 1 | 4 | 5
  Italy | 5 | 3 | 8
  Georgia | 1 | 1 | 2
  France | 3 | 3 | 6
  Serbia | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: PFS is defined as the time from randomization date until the date of disease progression, or death from any cause
Time Frame: 1 year 7 months
Population: A decision was made to terminate this Phase 3 study early due to business reasons. For the 82 subjects enrolled no scans had been collected at the time of termination, therefore no data were analyzed.
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of subjects who have a best overall response of CR or PR according to the Lugano Classification over the entire duration of the study, including the efficacy follow-up period.
Time Frame: 1 year 7 months
Population: as for outcome 1
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the proportion of subjects who have a best overall response of CR during the study (i.e., up to time of analysis of PFS).
Time Frame: 1 year 7 months
Population: A decision was made to terminate this Phase 3 study early due to business reasons. For the 84 subjects enrolled no scans had been collected at the time of termination, therefore no data were analyzed.
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Description: OS is defined as the time (in days) from randomization until death from any cause. For subjects alive at the time of analysis, they will be censored at the last documented alive date.
Time Frame: 1 year 7 months
Population: A decision was made to terminate this Phase 3 study early due to business reasons, therefore no data were collected or analyzed.
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Treatment Emergent AEs (Zandelisib When Combined With Rituximab)
Description: Measured by the number of Treatment Emergent AEs
Time Frame: 1 year 7 months
Population: Of the 41 subjects enrolled to the R+Zandelisib group 38 had a Treatment Emergent AE Of the 41 subjects enrolled to the R-Chemo group 37 had a Treatment Emergent AE
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Number analyzed (Participants) | 41 | 41
Participants | 38 | 37

6. Secondary Outcome: Number of SAEs (Zandelisib When Combined With Rituximab)
Description: Measured by the number of SAEs
Time Frame: 1 year 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Number analyzed (Participants) | 41 | 41
Participants | 12 | 8

7. Secondary Outcome: Number of Lab Abnormalities (Zandelisib When Combined With Rituximab)
Description: Measured by the number of laboratory abnormalities
Time Frame: 1 year 7 months
Population: A decision was made to terminate this Phase 3 study early due to business reasons. For the 82 subjects enrolled no lab abnormalities had been collected or analyzed
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The occurrence of adverse events was assessed for 1 year, 7 months
Description: 82 subjects were enrolled and dosed in the trial. 41 subjects in the Rituximab Zandelisib arm and in the R-chemo arm 31 subjects were assigned to R-B and 10 to R-CHOP.
Arm/Group | Rituximab Plus Zandelisib | Rituximab Plus Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/41 | 1/41
Serious Adverse Events (participants affected / at risk) | 12/41 | 8/41
Other Adverse Events (participants affected / at risk) | 38/41 | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Plus Zandelisib (N=41) | Rituximab Plus Chemotherapy (N=41)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Suspected Infection of unknown origin (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus Zandelisib (N=41) | Rituximab Plus Chemotherapy (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Corneal disorder (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 15 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 13
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 6
Asthenia (General disorders) | 2 | 2
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 2
Generalised oedema (General disorders) | 1 | 0
Injection site phlebitis (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 2
Mucosal inflammation (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 7
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 11 | 6
COVID-19 pneumonia (Infections and infestations) | 2 | 0
Candida infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 3 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Gastrointestinal fungal infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 1 | 0
Infected cyst (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Beta 2 microglobulin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 1
Cytomegalovirus test positive (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram QRS complex prolonged (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 3
Lymphocyte count increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 10 | 7
Platelet count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 2 | 2
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 3 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Presyncope (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 2 | 0
Suspected Infection of unknown origin (Infections and infestations) | 1 | 6
AST ALT increase (Investigations) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT04745832/Prot_002.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04745832/SAP_003.pdf